CLINICAL TRIAL: NCT04678648
Title: A Phase Ia/Ib, Open Label, Multi-center, Non-randomized Dose Escalation and Dose Expansion Study of RSC-1255 Alone or in Combination With Hydroxychloroquine in Patients With Advanced Solid Tumor Malignancies
Brief Title: A Trial of RSC-1255 for Treatment of Patients With Advanced Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: RasCal Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RSC-101
Record Dates: First submitted 2020-12-08; First posted 2020-12-22 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Advanced Malignant Solid Neoplasm; RAS Mutation; Lung Cancer; Colon Cancer; Glioblastoma; Pancreatic Cancer
Keywords: Malignancy; Cancer; Refractory; RAS mutation; Lung; Colon; Glioblastoma; RSC-1255; Progression; Pancreatic
MeSH Terms: conditions — Lung Neoplasms; Colonic Neoplasms; Glioblastoma; Pancreatic Neoplasms; Neoplasms; Disease Progression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- RSC-1255 Treatment (Experimental): Single Arm Study. All study participants receive RSC-1255.
  Interventions: Drug: RSC-1255 Dose Escalation; Drug: RSC-1255 Dose Expansion

INTERVENTIONS:
Drug: RSC-1255 Dose Escalation — Phase 1a will enroll 40-80 participants to identify the dose limiting toxicity (DLT), recommended Phase 1b dose, and the safety and tolerability of RSC-1255. RSC-1255 is administered orally twice daily, with and without food. Each cycle is 21 days.
  Other Names: Phase 1a; Dose Escalation
Drug: RSC-1255 Dose Expansion — Phase 1b will enroll 48-94 participants to further characterize the safety, pharmacology, and clinical efficacy of RSC-1255. RSC-1255 is administered orally twice daily alone or in combination with continuous hydroxychloroquine, with food. Each cycle is 21 days.
  Other Names: Phase 1b; Dose Expansion

SUMMARY:
RSC-101 is a Phase 1a/1b clinical trial of RSC-1255 in adult study participants with advanced solid tumor malignancies who are intolerant of existing therapies known to provide clinical benefit, have disease that has progressed after standard therapy, or have previously failed other therapies. The study has two phases. The purpose of Phase 1a (Dose Escalation) is to confirm the appropriate treatment dose and Phase 1b (Dose Expansion) is to characterize the safety and efficacy of RSC-1255.

DETAILED DESCRIPTION:
RSC-1255 is an orally bioavailable, small-molecule direct pan-mutant and wild-type RAS inhibitor. RSC-101 is a Phase 1a/1b, open-label, multi-center, non-randomized, Dose Escalation and Dose Expansion study in participants with advanced solid tumor malignancies. Study enrollment is approximately 134 participants. All participants receive oral RSC-1255, twice daily as monotherapy. Following Phase 1a (Dose Escalation) to identify the Maximum Tolerated Dose and Recommended Dose for use in Phase 1b, additional participants are enrolled in the Phase 1b (Dose Expansion) to further characterize the safety, pharmacology, and the clinical efficacy of RSC-1255 as monotherapy and in combination with the autophagy inhibitor hydroxychloroquine (HCQ).

ELIGIBILITY:
Inclusion Criteria (Key Factors):

1. Has pathologically confirmed advanced or metastatic malignancy characterized by one or more of the following:

   * Participant is intolerant of existing therapy(ies) known to provide clinical benefit for their condition
   * Malignancy is refractory to existing therapy(ies) known to potentially provide clinical benefit
   * Malignancy has progressed on standard therapy
2. Has evaluable or measurable tumor(s) in dose-escalation by standard radiological and/or laboratory assessments as applicable to their malignancy.
3. Has adequate performance status (PS): Eastern Co-operative Oncology Group (ECOG).
4. Is age ≥ 18 years.
5. Has either tissue agnostic tumors and documented RAS mutations or with glioblastoma with or without mutation in RAS

Exclusion Criteria (Key Factors):

1. Participants receiving cancer therapy at the time of enrollment.
2. Any clinically significant disease or condition affecting a major organ system.
3. Significant cardiovascular disease or electrocardiogram (ECG) abnormalities.
4. Known Gilbert's disease.
5. Has had a previous (within 2 years) or has a current malignancy other than the target cancer.
6. Intermittent hypokalemia
7. Grade 1 or higher nausea, vomiting, diarrhea at baseline due to underlying disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2021-03-03 (Actual); Primary Completion 2026-12-15 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) for RSC-1255 as monotherapy | Approximately 30 months
  The number and type of dose-limiting toxicities (DLTs) as defined in the protocol that occur during the first 21 days of treatment and maximum grade of all treatment-related events using CTCAE V5.0 will be used to identify a safe and tolerable dose.
Recommended Phase 2 Dose (RP2D) for RSC-1255 as monotherapy | Approximately 12 months
  The number and type of DLTs as defined in the protocol that occur during the first 21 days of treatment and maximum grade of all treatment-related adverse events using CTCAE 5.0 will be used to identify a safe and tolerable dose.

SECONDARY OUTCOMES:
Adverse event profile of RSC-1255 | Approximately 24 months
  Toxicities will be graded according to CTCAE V5.0.
Overall Survival (OS) | Approximately 24 months
  Overall Survival
Disease Progression | Approximately 24 months
  Disease Progression will be assessed using RECIST V1.1

CONTACTS AND LOCATIONS:
Overall Officials: Ali Manouchehri, MD, Study Director — RasCal Therapeutics, Inc.
Locations (3):
- United States (3):
  - University of California, Los Angeles (UCLA) Department of Medicine - Hematology/Oncology, Los Angeles, California
  - Sarah Cannon, SCRI Oncology Partners - Health One, Denver, Colorado
  - Sarah Cannon, SCRI Oncology Partners, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No